CLINICAL TRIAL: NCT05315726
Title: The Effects of Muscle Vibration on the Development of Spasticity and Neuroplasticity in a Post-stroke Population (Acute and Subacute Phases): Randomized Controlled Trial
Brief Title: The Effects of Muscle Vibration on the Development of Spasticity and Neuroplasticity in a Post-stroke Population
Acronym: SPACE-TIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JULLIAND AOIparaM 2021
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Post-stroke Patient in Acute, Sub-acute Phase or Chronic
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Muscle Strength Dynamometer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1 (Experimental)
  Interventions: Other: Dynamometer; Other: Muscle vibrations
- Phase 2: Intervention group (Experimental)
  Interventions: Other: Muscle vibrations
- Phase 2: control group (Active Comparator)
  Interventions: Other: Placebo muscle vibration

INTERVENTIONS:
Other: Dynamometer — Measurement of elbow/wrist spasticity
  Arms: Phase 1
Other: Muscle vibrations — 1 session of 10 minutes
  Arms: Phase 1
Other: Muscle vibrations — 3 times/week for 6 weeks
  Arms: Phase 2: Intervention group
Other: Placebo muscle vibration — 3 times/week for 6 weeks
  Arms: Phase 2: control group

SUMMARY:
Several studies have recently tested the use of muscle vibration for the rehabilitation of patients after a stroke. When applied in a repeated and focused manner, this vibration appears to promote the recovery of functional capacities through the mechanisms of neuromuscular plasticity. These results are encouraging, showing in particular a significant decrease in spasticity in post-stroke patients in the chronic phase (> 6 months after stroke), on the upper and/or lower limbs. However, very few studies have been done on this type of early intervention. Muscle vibration may therefore be an innovative therapy to complement the care that is currently offered in the acute and subacute phase of post-stroke rehabilitation.

Moreover, brain plasticity after a stroke is particularly high in the 3 months after the accident, but the vast majority of studies having evaluated the impact of vibration in a chronic phase (> 12 months post-stroke). It is likely, however, that the influence of vibration, particularly on brain plasticity, is increased in the acute or subacute phase (first 6 months). To date, the effect of vibration on spinal cord or cortical plasticity has not been quantified in the acute or subacute phase. This is why the second part of this project (phase 2) aims to systematically evaluate and quantify the neuroplastic and functional effects of post-stroke vibration in the early phase.

Phase 1 - Validation of a method for measuring spasticity (upper limb) with an isokinetic dynamometer 32 patients with ischemic and/or hemorrhagic stroke (> 3 months after stroke)

Phase 2 - Use of this objective technique to measure the effect of a muscle vibration protocol to limit the onset of spasticity in a population of 100 patients following a stroke, in the acute or subacute phase (< 6 weeks post-stroke) in a randomized trial:

* intervention group: usual rehabilitation + muscle vibrations
* control group: usual rehabilitation + placebo vibrations

ELIGIBILITY:
Inclusion Criteria:

Phase 1:

* Adult patient,
* Medically stable on medical assessment, with no contraindications to stroke rehabilitation management management (no medical problems or acute intercurrent medical events),
* Have had an ischemic and/or hemorrhagic stroke (> 3 months post-stroke), impacting the motor skills of the upper limbs,
* 1 ≤ MAS < 4 on elbow or wrist flexors,
* Having given oral consent.

Phase 2:

* Adult patient > 18 years old,
* Able to follow a rehabilitation program on medical opinion (no medical issues or acute intercurrent medical events),
* First stroke ever < 6 weeks, confirmed by imaging,
* Hemiparesis or hemiplegia of the upper limb (FMA-UE score < 48), particularly in the wrist and elbow flexors,
* Requiring inpatient or outpatient hospitalization in a rehabilitation center,
* Having given oral consent.

Exclusion Criteria:

* Phases 1 and 2:
* Significant pain on mobilization of the wrist or elbow (VAS > 5/10),
* Presence of other neurological, muscular or osteoarticular conditions altering upper limb function,
* Apparent wound, which may postpone inclusion, or very fragile skin,
* Significant cognitive impairments: inability to understand simple instructions or give consent of any kind (not included if: LAST scores < 5/7 in comprehension, and if YES/NO answers are unreliable),
* Not covered by national health insurance,
* Being pregnant or breastfeeding,
* Being under guardianship or curatorship.
* Person subject to a measure of legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Joint angle (elbow or wrist of the limb contralateral to the brain injury) | at baseline
  Joint angle (elbow or wrist of the limb contralateral to the brain injury) at the onset of a spastic contraction (maximum intensity of resistance to mobilization) recorded by isokinetic dynamometer on a wheelchair during the initial visit
Phase 2: Scoring wrist flexor muscle spasticity | at 6 weeks
  Scoring of wrist flexor muscle spasticity by the Modified Ashworth Scale (MAS), at the beginning of the study and at 6 weeks (end of intervention).

SECONDARY OUTCOMES:
Sensorimotor function modifications of the paretic upper limb | at 0, 6 weeks and 6 months
  Fugl-Meyer Assessment of Upper Extremity (FMA-UE)
Sensorimotor function modifications of the paretic upper limb | at 0, 6 weeks and 6 months
  Pain (Visual analog scale)
Sensorimotor function modifications of the paretic upper limb | at 0, 6 weeks and 6 months
  tiredness (Visual analog scale)
Spasticity of the paretic limb at the wrist | at 0, 3 weeks, 6 weeks and 6 months
  Angle of catch of spasticity measured by an isokinetic ergometer (in degree), only in Dijon
Spasticity of the paretic limb at the wrist | at 0, 3 weeks, 6 weeks and 6 months
  Angle of end of spasticity measured by an isokinetic ergometer (in degree), only in Dijon
Spasticity of the paretic limb at the wrist | at 0, 3 weeks, 6 weeks and 6 months
  Measured by an isokinetic ergometer : Torque developed during the spastic reaction that is determined by the angles of catch and end (in Newton per Meter (Nm)). It will be reported as a score difference in comparison to the reference curve: root mean square error (RMSE) only in Dijon
Spasticity of the paretic limb at the elbow | at 0, 3 weeks, 6 weeks and 6 months
  Angle of catch of spasticity measured by an isokinetic ergometer (in degree), only in Dijon
Spasticity of the paretic limb at the elbow | at 0, 3 weeks, 6 weeks and 6 months
  Angle of end of spasticity measured by an isokinetic ergometer (in degree), only in Dijon
Spasticity of the paretic limb at the elbow | at 0, 3 weeks, 6 weeks and 6 months
  Measured by an isokinetic ergometer : Torque developed during the spastic reaction that is determined by the angles of catch and end (in Newton per Meter (Nm)). It will be reported as a score difference in comparison to the reference curve: root mean square error (RMSE) only in Dijon
Spasticity of the paretic limb (wrist and elbow) | at 0, 3 weeks, 6 weeks and 6 months
  Measured by the Modified Ashworth Scale (MAS)
Neuroplasticity modifications evaluated on the flexor carpi radialis | at 0, 3 weeks, 6 weeks and 6 months
  at spinal level (H-reflex and M-wave), Only in Dijon.
Neuroplasticity modifications evaluated on the flexor carpi radialis | at 0, 3 weeks, 6 weeks and 6 months
  at corticospinal level by transcranial magnetic stimulation (MEP and SICI), Only in Dijon.
Neuroplasticity modifications evaluated on the flexor carpi radialis | at 0, 3 weeks, 6 weeks and 6 months
  at cortical level by electroencephalogram : The Delta, Theta, Alpha and Beta bands will be evaluated. ERD/ERS will be calculated during the resting states and the vibrations periods, principally over the C3-C4 electrodes (10-20 system).
  Only in Dijon.
Correlation between the severity of spasticity at the wrist and the spinal excitability | Through study completion, on average of 6 months
  Tools: MAS scores (scale) and the amplitude of the H-reflex (in Volt) Logistic regression Only in Dijon.
Correlation between the severity of spasticity at the wrist and cortical excitability | Through study completion, on average of 6 months
  Tools: MAS scores (scale) and EEG ratio (laterality coefficient) Logistic regression Only in Dijon.
Correlation between the severity of spasticity at the wrist and cortical excitability | Through study completion, on average of 6 months
  Tools: MAS scores (scale) and EEG ratio (ERD alpha and beta bands) Logistic regression Only in Dijon.
Correlation between the severity of spasticity at the wrist and the spinal excitability | Through study completion, on average of 6 months
  Tools: Angle of catch (in degree) and the amplitude of the H-reflex (in Volt) Logistic regression Only in Dijon.
Correlation between the severity of spasticity at the wrist and cortical excitability | Through study completion, on average of 6 months
  Tools: Angle of catch (in degree) and EEG ratio (laterality coefficient) Logistic regression Only in Dijon.
Correlation between the severity of spasticity at the wrist and cortical excitability | Through study completion, on average of 6 months
  Tools: Angle of catch (in degree) and EEG ratio (ERD alpha and beta bands)) Logistic regression Only in Dijon.
Correlation between the severity of spasticity at the wrist and the spinal excitability | Through study completion, on average of 6 months
  Tools: Torque score (RMSE) and the amplitude of the H-reflex (in Volt) Logistic regression Only in Dijon.
Correlation between the severity of spasticity at the wrist and cortical excitability | Through study completion, on average of 6 months
  Tools: Torque score (RMSE) and EEG ratio (laterality coefficient) Logistic regression Only in Dijon
Correlation between the severity of spasticity at the wrist and cortical excitability | Through study completion, on average of 6 months
  Tools: Torque score (RMSE) and EEG ratio (ERD alpha and beta bands)) Logistic regression Only in Dijon

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - SSR Marguerite BOUCICAUT, Chalon-sur-Saône
  - Chu Dijon Bourgogne, Dijon

IPD SHARING:
Plan to Share IPD: Yes
The study team policy is about to share and collaborate with other research teams upon reasonable request for access to study data. Expressions of interest in access to study data, addressed to the corresponding author, will be considered and data de-identified at group or individual level may be shared as appropriate. A data transfer agreement will then be drawn up. The study dataset will be available at the end of the study, once the database is frozen. Sharing the database will be made available between interested parts with a data sharing agreement contract.
Supporting Information: Analytic Code
Time Frame: after publication of the lead article

REFERENCES:
- [Derived] Julliand S, Papaxanthis C, Delphin C, Mock A, Raumel MA, Gueugnon M, Ornetti P, Laroche D. IMPROVE study protocol, investigating post-stroke local muscle vibrations to promote cerebral plasticity and functional recovery: a single-blind randomised controlled trial. BMJ Open. 2024 Mar 15;14(3):e079918. doi: 10.1136/bmjopen-2023-079918. PMID 38490651